CLINICAL TRIAL: NCT01677975
Title: The Value of Preoperative Dynamic Lymphscintigraphy and Ultrasoundscanning, Eventually With FNA, for Identification of Malignant Sentinel Node(s) in Patients With Melanoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Trine-Lise Lambine, afdelingslæge, Rigshospitalet, Denmark
Other Study IDs: Ultrasound in melanomas
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultrasound, dynamic lymphscintigraphy (Experimental)
  Interventions: Procedure: FNA (fine needle aspiration)

INTERVENTIONS:
Procedure: FNA (fine needle aspiration)

SUMMARY:
The goal with this study is to evaluate the value of dynamic lymphscintigraphy and ultrasoundscanning preoperative in patients with melanomas.

ELIGIBILITY:
Inclusion Criteria:

Histologically verified melanomas, at least 1 mm thickness, or thinner melanomas with ulceration and/or Clarks level IV-V and/or mitoserate at least 1/mm2.

Exclusion Criteria:

Other malignant illness Known local, regional or non-regional metastasis on the time of diagnonsis Comorbidity which contraindicate lymphnoderemoval Age less than 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-09

CONTACTS AND LOCATIONS:
Locations (1):
- Ultrasounddepartment 4123, Rigshospitalet, Blegdamsvej 9, København Ø, Denmark